CLINICAL TRIAL: NCT02371902
Title: Extracorporeal Shock Wave Therapy vs Cryoultrasound Therapy in the Treatment of Chronic Lateral Epicondylitis: One Year Follow up Study
Brief Title: ESWT vs Cryo-US Therapy in the Treatment of Chronic Lateral Epicondylitis: One Year Follow up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mario Vetrano, MD, MD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-02-12; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Tendinopathy
Keywords: Elbow pain; lateral epicondylitis; conservative treatment; shock wave treatment; therapeutic ultrasound
MeSH Terms: conditions — Tendinopathy; Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESWT Group (Active Comparator): Focused Extracorporeal Shock Wave Therapy: 3 sessions were carried out, with the time interval between sessions spanning between 48 and 72 hours. In each session, 2400 pulses were administered with energy flux density (EDF) ranging from 0.14 and 0.20 mJ/mm2
  Interventions: Device: MODULITH® SLK, STORZ MEDICAL AG, Switzerland
- Cryo-US Group (Active Comparator): Therapeutic cryoultrasound: 12 sessions was performed in a continuous emission modality, using an ultrasound emission power rating of 1,8 Watt/cm2, and a temperature of -2˚C, for a total of 12 sessions lasting 20 minutes each.
  Interventions: Device: Cryoultrasound™, Medisport S.r.l., Italy

INTERVENTIONS:
Device: MODULITH® SLK, STORZ MEDICAL AG, Switzerland — Three sessions were carried out, with the time interval between sessions spanning between 48 and 72 hours. In each session, 2400 pulses were administered with energy flux density (EDF) ranging from 0.14 and 0.20 mJ/mm2, depending on the maximum tolerated pain of each patient. Analgesics or local anaesthetics were not administered before, during or after treatment.
  Other Names: Focused Extracorporeal Shock Wave Therapy; ESWT
  Arms: ESWT Group
Device: Cryoultrasound™, Medisport S.r.l., Italy — Cryo-US therapy was performed in a continuous emission modality, using an ultrasound emission power rating of 1,8 Watt/cm2, and a temperature of -2˚C, for a total of 12 sessions lasting 20 minutes each. The treatment was performed in 3 weeks (4 daily sessions per week).
  Other Names: Therapeutic Ultrasound; Cryo-US therapy
  Arms: Cryo-US Group

SUMMARY:
Chronic lateral epicondylitis is usually managed conservatively. The purpose of this single-blinded, randomized, controlled study is to compare the clinical therapeutic effects of extracorporeal shock wave therapy (ESWT) in comparison with cryoultrasound (Cryo-US) therapy in chronic lateral epicondylitis (LE) during a period of 12 months.

DETAILED DESCRIPTION:
Eighty participants with chronic LE were randomly assigned to receive 3 ESWT sessions at 48/72-hours intervals -2400 impulses at energy flux density 0.14-0.20 mJ/mm2 at each session- (ESWT Group, n=40) or 12 Cryo-US therapy sessions (4 daily sessions per week) in a continuous modality at 1.8 Watt/cm2 and -2˚C at each session- (Cryo-US Group, n=40). Visual Analogue Scale (VAS) and satisfactory results, considered as the sum of the excellent and good scores in the Roles and Maudsley score, were used as outcome measures at baseline and 3, 6, and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* an age range from 18 to 75 years
* clinical or instrumental diagnosis of chronic lateral epicondylitis, present for at least three months
* intensity of pain of more than 5 on the Visual Analogue Scale (VAS) performing a maximum voluntary resisted isometric wrist extension with the elbow in extension (Cozen test)
* the failure of conservative treatments previously made
* a wash-out period of at least 12 weeks since the last conservative therapy carried out before inclusion in the study
* capability of filling in the questionnaires and signing the consent form

Exclusion Criteria:

* Previous treatment with Cryo-US, ultrasound therapy, ESWT
* The conjoint presence of bilateral or lateral and medial epicondylitis
* Acute infection of the soft tissues or the bones adjacent to the area of treatment
* Local bleedings or skin lesions, pathologies of the blood coagulation, or use of anticoagulant drugs
* Pacemaker, pregnancy
* Neoplastic disease
* Raynaud's disease, altered thermal and pain sensitivity, or cold intolerance
* Evidence of elbow bursitis, or articular or synovial pathologies; signs of elbow laxity or instability
* Cervicobrachialgia; syndrome of ulnar, radial, or posterior interosseous nerve entrapment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Difference of two points in pain recorded on the VAS | 3, 6, or 12 months after the end of treatments
  a difference of two points in pain recorded on the VAS during a maximum voluntary resisted isometric wrist extension with the elbow in extension (Cozen test), between the ESWT Group and the Cryo-US Group, in at least one of the periods taken into account.

SECONDARY OUTCOMES:
Patients satisfaction based on the Roles and Maudsley score | 3, 6, or 12 months after the end of treatments
  the number of patients who achieved at least 50% satisfactory results at 3, 6 and 12 months after the treatment. Satisfactory results were described as the sum of the excellent and good scores based on the Roles and Maudsley score.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Vulpiani, MD, Study Chair — La Sapienza University of Rome
Locations (1):
- Sant'Andrea Hospital, Rome, Italy, Italy

REFERENCES:
- [Result] Shiri R, Viikari-Juntura E, Varonen H, Heliovaara M. Prevalence and determinants of lateral and medial epicondylitis: a population study. Am J Epidemiol. 2006 Dec 1;164(11):1065-74. doi: 10.1093/aje/kwj325. Epub 2006 Sep 12. PMID 16968862
- [Result] Kraushaar BS, Nirschl RP. Tendinosis of the elbow (tennis elbow). Clinical features and findings of histological, immunohistochemical, and electron microscopy studies. J Bone Joint Surg Am. 1999 Feb;81(2):259-78. No abstract available. PMID 10073590
- [Result] Galloway MT, Lalley AL, Shearn JT. The role of mechanical loading in tendon development, maintenance, injury, and repair. J Bone Joint Surg Am. 2013 Sep 4;95(17):1620-8. doi: 10.2106/JBJS.L.01004. PMID 24005204
- [Result] Haahr JP, Andersen JH. Prognostic factors in lateral epicondylitis: a randomized trial with one-year follow-up in 266 new cases treated with minimal occupational intervention or the usual approach in general practice. Rheumatology (Oxford). 2003 Oct;42(10):1216-25. doi: 10.1093/rheumatology/keg360. Epub 2003 Jun 16. PMID 12810936
- [Result] Dingemanse R, Randsdorp M, Koes BW, Huisstede BM. Evidence for the effectiveness of electrophysical modalities for treatment of medial and lateral epicondylitis: a systematic review. Br J Sports Med. 2014 Jun;48(12):957-65. doi: 10.1136/bjsports-2012-091513. Epub 2013 Jan 18. PMID 23335238
- [Result] Vetrano M, d'Alessandro F, Torrisi MR, Ferretti A, Vulpiani MC, Visco V. Extracorporeal shock wave therapy promotes cell proliferation and collagen synthesis of primary cultured human tenocytes. Knee Surg Sports Traumatol Arthrosc. 2011 Dec;19(12):2159-68. doi: 10.1007/s00167-011-1534-9. Epub 2011 May 27. PMID 21617986
- [Result] Leone L, Vetrano M, Ranieri D, Raffa S, Vulpiani MC, Ferretti A, Torrisi MR, Visco V. Extracorporeal Shock Wave Treatment (ESWT) improves in vitro functional activities of ruptured human tendon-derived tenocytes. PLoS One. 2012;7(11):e49759. doi: 10.1371/journal.pone.0049759. Epub 2012 Nov 26. PMID 23189160
- [Result] Speed CA. Therapeutic ultrasound in soft tissue lesions. Rheumatology (Oxford). 2001 Dec;40(12):1331-6. doi: 10.1093/rheumatology/40.12.1331. PMID 11752501
- [Result] Tsai WC, Pang JH, Hsu CC, Chu NK, Lin MS, Hu CF. Ultrasound stimulation of types I and III collagen expression of tendon cell and upregulation of transforming growth factor beta. J Orthop Res. 2006 Jun;24(6):1310-6. doi: 10.1002/jor.20130. PMID 16705693
- [Result] Costantino C, Pogliacomi F, Vaienti E. Cryoultrasound therapy and tendonitis in athletes: a comparative evaluation versus laser CO2 and t.e.ca.r. therapy. Acta Biomed. 2005 Apr;76(1):37-41. PMID 16116824
- [Result] Costantino C, Vulpiani MC, Romiti D, Vetrano M, Saraceni VM. Cryoultrasound therapy in the treatment of chronic plantar fasciitis with heel spurs. A randomized controlled clinical study. Eur J Phys Rehabil Med. 2014 Feb;50(1):39-47. Epub 2013 Oct 30. PMID 24172641
- [Result] Chung B, Wiley JP, Rose MS. Long-term effectiveness of extracorporeal shockwave therapy in the treatment of previously untreated lateral epicondylitis. Clin J Sport Med. 2005 Sep;15(5):305-12. doi: 10.1097/01.jsm.0000179137.69598.7e. PMID 16162988
- [Result] Radwan YA, ElSobhi G, Badawy WS, Reda A, Khalid S. Resistant tennis elbow: shock-wave therapy versus percutaneous tenotomy. Int Orthop. 2008 Oct;32(5):671-7. doi: 10.1007/s00264-007-0379-9. Epub 2007 Jun 6. PMID 17551726
- [Result] Rompe JD, Decking J, Schoellner C, Theis C. Repetitive low-energy shock wave treatment for chronic lateral epicondylitis in tennis players. Am J Sports Med. 2004 Apr-May;32(3):734-43. doi: 10.1177/0363546503261697. PMID 15090392
- [Result] Day B. 'Extracorporeal shock wave therapy for lateral epicondylitis--a double blind randomised controlled trial', by Speed CA, Nichols D, Richards C, Humphreys H, Wies JT, Burnet S, Hazleman BL [Journal of Orthopaedic Research 29 (2002) 895-898]. J Orthop Res. 2003 Sep;21(5):960; author reply 961. doi: 10.1016/S0736-0266(03)00045-7. No abstract available. PMID 12919888
- [Result] Rompe JD, Overend TJ, MacDermid JC. Validation of the Patient-rated Tennis Elbow Evaluation Questionnaire. J Hand Ther. 2007 Jan-Mar;20(1):3-10; quiz 11. doi: 10.1197/j.jht.2006.10.003. PMID 17254903